CLINICAL TRIAL: NCT01303315
Title: TANTALUS Therapy in Type 2 Diabetic Patients Intolerant or Inadequately Responsive to GLP-1 Receptor Agonist Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company strategic decision
Sponsor: MetaCure (USA), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC CPTAN2010-017; Position II (Other: MetaCure)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: C19 246 300
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GLP-1 receptor agonist therapy (Other): Group A: Subjects on GLP-1 receptor agonist therapy only. After run in of 12 weeks on GLP-1 receptor agonist therapy, Patients with HbA1c < 7.5 are moved to Group A, continue GLP-1 receptor agonist therapy, and then start the Evaluation Period These patients will not be implanted with the TANTALUS system.
  Interventions: Device: TANTALUS System
- GLP-1 receptor agonist and TANTALUS (Experimental): Group B: subjects on GLP-1 receptor agonist therapy and TANTALUS therapy After run in of 12 weeks on GLP-1 receptor agonist therapy, Patients with HbA1c > 7.5 are moved to Group B, continue GLP-1 receptor agonist therapy, implanted with TANTALUS within 4 weeks, and then start the Evaluation Period
  Interventions: Device: TANTALUS System
- Subjects on TANTALUS therapy only (Active Comparator): Group C: subjects on TANTALUS therapy only After run in of 12 weeks on GLP-1 receptor agonist therapy, patients intolerant to low dosage of GLP-1 receptor agonist therapy will be implanted with the TANTALUS system
  Interventions: Device: TANTALUS System

INTERVENTIONS:
Device: TANTALUS System — An Active Implantable Pulse Generator Medical Device for the treatment of Obesity and Diabetes Type 2 and Obesity
  Other Names: TANTALUS System, TANTALUS II

SUMMARY:
To assess the TANTALUS therapy in type 2 diabetic patients who can not tolerate GLP-1 agonist due to unacceptable side effects; and to assess the TANTALUS therapy in type 2 diabetic patients who do not sufficiently benefit from GLP-1 receptor agonist therapy

DETAILED DESCRIPTION:
The present protocol will address whether the effects of the TANTALUS treatment are complimentary to GLP-1 treatment which is only partially effective or whether it can replace GLP-1 treatment in individuals who cannot tolerate GLP-1 agonists because of unacceptable side effects.

This investigation will be a 3 arm multicenter study which will enroll in a Run-In Period up to 400 with type 2 diabetes mellitus. This Run-In Period will facilitate screening the patients with the aim to have a maximum of 30 patients in each arm complete the Evaluation Period of 6 months. The study aims at evaluating the TANTALUS therapy compared to GLP-1 receptor agonist therapy by evaluating improvement in glycemic control and weight after 6 months of treatment in each of the 3 study groups, which are:

* Group A: subjects on GLP-1 receptor agonist therapy only
* Group B: subjects on GLP-1 receptor agonist therapy and TANTALUS therapy
* Group C: subjects on TANTALUS therapy only

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 21 through 70 years of age
2. Type 2 diabetes duration more than 6 months and less than 10 years
3. 7.8% < HbA1c < 10.5% if T2DM duration less than or equal to 5 years
4. 7.8% < HbA1c < 10.0% if T2DM duration more than 5 years
5. BMI < 40 kg/m2
6. Taking at least one oral anti-diabetic medication
7. Patients treated with GLP-1 receptor agonist with at least one oral anti-diabetic medication may be included under the following conditions:

   a. The HbA1c, before GLP-1 receptor agonist therapy was administered, was: i. 7.8% < HbA1c < 10.5% if T2DM duration less than 5 years ii. 7.8% < HbA1c < 10.0% if T2DM duration greater than 5 years b. The patient was on GLP-1 receptor agonist therapy for no more than 12 weeks
8. Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods
9. If subject is taking lipid-lowering medication, the treatment must be stable for at least one month prior to enrollment
10. If subject is taking anti-hypertensive medication, the treatment must be stable for at least one month prior to enrollment
11. If subject is taking anti-depressant medication, the treatment must be stable for at least one month prior to enrollment
12. Willingness to refrain from using prescription, over the counter, or herbal weight loss products for the duration of the trial
13. Ability and willingness to perform required study and data collection procedures and adhere to operating requirements of the TANTALUS® System
14. Alert, mentally competent, and able to understand and willing to comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial
15. Able to provide voluntary informed consent

Exclusion Criteria:

1. Insulin therapy within the last 3 months 2. GLP-1 receptor agonist therapy longer than 3 months 3. Diagnosed with renal dysfunction or history of renal dysfunction 4. Taking medications known to affect gastric motility 5. Use of prescription, over the counter or herbal weight loss products or obesity drugs during the past two months 6. Experiencing severe and progressing diabetic complications (7. Prior wound healing problems 8. Diagnosed with past or current psychiatric condition that may impair his or her ability to comply with the study procedures 9. Use of anti-psychotic medications 10. Diagnosed with eating disorder such as bulimia or binge eating 11. Obesity due to an endocrinopathy 12. Hiatal hernia requiring surgical repair or a paraesophageal hernia 13. Pregnant or lactating 14. Diagnosed with impaired liver function 15. Any prior bariatric surgery 16. Any history of pancreatitis 17. Any history of peptic ulcer disease within 5 years of enrollment 18. Diagnosed with Gastroparesis or other GI motility disorder 19. Use of active medical devices (either implantable or external) such as ICD, drug infusion device, or neurostimulator (either implanted or worn). Subjects using an external active device who are able and willing to avoid use of the device during the study may be enrolled.

20. Cardiac history that physician feels should exclude the subject from the study.

21. Use of another investigational device or agent in the 30 days prior to enrollment 22. A history of life-threatening disease within 5 years of enrollment 23. Any additional condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Decrees in HbA1c of at least 0.5 points and Weight loss of at least 3% of total body weight after 6 month of treatment | 6 month
  Change in HbA1c and weight will be assessed at baseline and 24 weeks of treatment for Group A and C.
  Additionally, each group will be analyzed for the weight of decrease extent, the percentage of patients achieving the endpoint, and the percentage of patients that reach an HbA1c less than 7.0%.

SECONDARY OUTCOMES:
Glycemic and metabolic parameters | 6 month
  * Glycemic Parameters (FBG, PPG)
  * Glycemic Dynamics (Glucose, Insulin, C-Peptide, and Glucagon Profiles) via MTT
  * Metabolic Parameters (WC, BP, Lipids, Gastric Emptying)
  * Gastric Hormones (GLP-1, GIP, Ghrelin, PYY, Pancreatic Polypeptide) via MTT

CONTACTS AND LOCATIONS:
Overall Officials: Walid Haddad, PhD, Study Director — MetaCure Limited
Locations (13):
- Czechia (4):
  - Fakultni Nemocnice U SV. Anny V Brne, Brno
  - Klinika gerontologická a metabolická,, Hradec Králové
  - General University Hospital,, Prague
  - Prednosta OB Kliniky a.s.,, Prague
- Germany (3):
  - Asklepios Klinik St. Georg, Hamburg, Hamburg
  - Diabetes Zentrum, Bad Mergentheim
  - Diabetes-Praxis Muenster, Münster
- Romania (6):
  - 'N. Paulescu' National Institute of Diabetes, Nutrition and Metabolic Diseases, Bucharest
  - CMI Dr Busegeanu Mihaela Magdalena-Ploiesti, Bucharest
  - Fundeni Hospital - Surgical, Bucharest
  - Sanatatea Ta Medical Center, Bucharest
  - Sf. Ioan Hospital - Surgical, Bucharest
  - Spitalul Pelican, Orada, Bucharest